CLINICAL TRIAL: NCT00450801
Title: Phase II Study of Rituximab in Combination With Methotrexate, Doxorubicin, Cyclophosphamide, Leucovorin, Vincristine, Ifosfamide, Etoposide, Cytarabine and Mesna (MACLO/IVAM) in Patients With Previously Untreated Mantle Cell Lymphoma
Brief Title: R-MACLO-IVAM and Thalidomide in Untreated Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Izidore Lossos, Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20030165; SCCC-2003027 (Other: University of Miami Sylvester Comprehensive Cancer Center); WIRB-20051242 (Other: Western Institutional Review Board)
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Results first posted 2015-11-10 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-10

CONDITIONS: Lymphoma
Keywords: contiguous stage II mantle cell lymphoma; noncontiguous stage II mantle cell lymphoma; stage I mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell | interventions — Rituximab; Cyclophosphamide; Cytarabine; Doxorubicin; Etoposide; Ifosfamide; Leucovorin; Methotrexate; Thalidomide; Vincristine; Mesna; Filgrastim; Granulocyte Colony-Stimulating Factor; Granisetron; Calcium Dobesilate; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- R-MACLO-IVAM-T (Experimental): Rituximab, Methotrexate, Doxorubicin, Cyclophosphamide and Vincristine (cycle 1), followed by Rituximab, Ifosfamide (and Mesna), Etoposide and Cytarabine (cycle 2). These two cycles are repeated once, and patients achieving complete repose receive maintenance Thalidomide.
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Doxorubicin; Drug: Etoposide; Drug: Ifosfamide; Drug: Leucovorin; Drug: Methotrexate; Drug: Thalidomide; Drug: Vincristine; Drug: Mesna; Drug: Filgrastim (G-CSF); Drug: Granisetron; Drug: Decadron

INTERVENTIONS:
Drug: Rituximab — Rituximab 375 mg/m2 IV, Days 1 of all cycles
  Other Names: Rituxan
Drug: Cyclophosphamide — Cyclophosphamide 800 mg/m2 IV, Day 1, Cyclophosphamide 200 mg/m2 IV Days 2 - 5, Cycles 1 and 3. Cyclophosphamide will be given in 100 cc NS IV over 30 minutes.
  Other Names: Cytoxan
Drug: Cytarabine — Cytarabine 2 grams/m2 IV every 12 hours x 4 doses, Days 1 and 2, Cycles 2 and 4.
  Other Names: AraC
Drug: Doxorubicin — Doxorubicin 45 mg/m2 IV bolus, Day 1, Cycles 1 and 3
  Other Names: Adriamycin
Drug: Etoposide — Etoposide 60 mg/m2 IV daily x 5 days, Cycles 2 and 4
  Other Names: VP16
Drug: Ifosfamide — Ifosfamide 1.5 grams/m2 IV once a day (QD) x 5 days, Cycles 2 and 4
  Other Names: Ifex
Drug: Leucovorin — Leucovorin 180 mg/m2 IV beginning 36 hours after start of methotrexate infusion and then 12 mg/m2 IV every 6 hours until methotrexate level is below 0.01 nM. Day 10, Cycles 1 and 3.
  Other Names: Folinic Acid
Drug: Methotrexate — Methotrexate 1,200 mg/m2 in 250 cc 5 percent dextrose in water (D5W) IV over 1 hour followed by Methotrexate 5,520 mg/m2 in 1,000 cc D5W by continuous infusion over 23 hours (240 mg/m2 every hour for 23 hours). Day 10, Cycles 1 and 3.
  Other Names: amethopterin
Drug: Thalidomide — Maintenance therapy.
  Other Names: Thalomid
Drug: Vincristine — Vincristine 1.5 mg/m2 IVP (maximum of 2 mg), Day 1 and 8 , Cycles 1 and 3.
  Other Names: Oncovin
Drug: Mesna — Mesna 360 mg/m2 IV every 3 hours x 5 days, Cycles 2 and 4
  Other Names: Mesnex
Drug: Filgrastim (G-CSF) — G-CSF 480 mcg subcutaneous (SQ) starting Day 13 (Cycles 1 and 3), Day 7 (Cycles 2 and 4)
  Other Names: Neupogen
Drug: Granisetron — Granisetron 1 mg IV on Day 1, Cycle 1 and 3
  Other Names: Sancuso; Granisol
Drug: Decadron — Decadron 10 mg IV on Day 1, Cycles 1 and 3
  Other Names: Maxidex; Ozurdex; Baycadron

SUMMARY:
RATIONALE: To evaluate the efficacy of a new high intensity chemotherapy regimen with thalidomide maintenance in patients with newly diagnosed mantle cell lymphoma

PURPOSE: This phase II trial is studying how well giving rituximab together with combination chemotherapy followed by thalidomide works in treating patients with previously untreated mantle cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the progression-free survival of patients with previously untreated mantle cell lymphoma treated rituximab in combination with methotrexate, doxorubicin, cyclophosphamide, leucovorin, vincristine, ifosfamide, etoposide, cytarabine and mesna (MACLO/IVAM) followed by thalidomide.

Secondary

* Determine the overall survival of patients treated with this regimen.
* Determine the response rate in patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.

OUTLINE: During cycle 1, patients will receive rituximab intravenous (IV), granisetron IV, decadron IV, doxorubicin IV bolus, vincristine intravenous pyelogram (IVP) on day 1; cyclophosphamide IV on day 1-5; vincristine IVP on day 8; methotrexate IV, methotrexate by continuous infusion, then leucovorin IV until methotrexate level is below 0.01 nanomolar (nM) on day 10. Patients will receive filgrastim (G-CSF) subcutaneously (SC) once daily beginning on day 13 and continuing until blood counts recover.

When absolute neutrophil count (ANC) reaches1,500/mm^3, patients will start cycle 2. Patients will receive rituximab IV on day 1; cytarabine IV on day 1 and 2; ifosfamide IV, mesna IV, etoposide IV on day 1-5; and G-CSF SC daily beginning on day 7 and continuing until ANC is greater than 1,000 cells/mm^3.

Approximately 2-3 weeks later, patients receive another course of therapy as above.After cycle 4, patients in complete remission will take oral thalidomide until progression of disease. After completion of study treatment, patients are followed monthly for 3 months, every 3 months for 2 years, every 6 months for 3-5 years, and then annually thereafter or at study termination.

PROJECTED ACCRUAL: A total of 22 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated, histologically confirmed mantle cell lymphoma.
* Measurable or evaluable disease.
* All stages are eligible.
* Age > 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2.
* Adequate hepatic function:

  * Bilirubin < 3 mg/dL.
  * Transaminases (SGOT and/or SGPT) < than 2.5 times the upper limit of normal for the institution, unless due to lymphomatous involvement.
* Serum creatinine < 1.5 mg/Dl.
* Ability to give informed consent.
* Women of childbearing potential must have a negative pregnancy test within 72 hours of entering into the study. Males and females must agree to use adequate birth control if conception is possible during the study. Women must avoid pregnancy and men avoid fathering children while in the study.
* Life expectancy greater than 6 months.

Exclusion Criteria:

* Previous chemotherapy, immunotherapy or radiotherapy for this lymphoma
* Concurrent active malignancies, with the exception of in situ carcinoma of the cervix and basal cell carcinoma of the skin.
* Grade 3 or 4 cardiac failure and/or ejection fraction < 50.
* Psychological, familial, sociological or geographical conditions that do not permit treatment and/or medical follow-up required to comply with the study protocol.
* Patients with a known history of HIV or AIDS
* Presence of hepatitis or hepatitis B virus (HBV) infection
* Pregnant or breast-feeding women.
* Central nervous system (CNS) involvement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2004-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Izidore S. Lossos, MD, Study Chair — University of Miami Sylvester Comprehensive Cancer Center
Locations (1):
- University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida, United States

REFERENCES:
- [Result] Lossos IS, Hosein PJ, Morgensztern D, Coleman F, Escalon MP, Byrne GE Jr, Rosenblatt JD, Walker GR. High rate and prolonged duration of complete remissions induced by rituximab, methotrexate, doxorubicin, cyclophosphamide, vincristine, ifosfamide, etoposide, cytarabine, and thalidomide (R-MACLO-IVAM-T), a modification of the National Cancer Institute 89-C-41 regimen, in patients with newly diagnosed mantle cell lymphoma. Leuk Lymphoma. 2010 Mar;51(3):406-14. doi: 10.3109/10428190903518345. PMID 20038221
- [Derived] Alderuccio JP, Saul EE, Iyer SG, Reis IM, Alencar AJ, Rosenblatt JD, Lossos IS. R-MACLO-IVAM regimen followed by maintenance therapy induces durable remissions in untreated mantle cell lymphoma - Long term follow up results. Am J Hematol. 2021 Jun 1;96(6):680-689. doi: 10.1002/ajh.26163. Epub 2021 Apr 7. PMID 33735476

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | R-MACLO-IVAM-T
Started | 22
Completed | 21
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | R-MACLO-IVAM-T
Number analyzed (Participants) | 22
Age, Continuous [Median (Full Range); unit: years] | 56.5 [39 to 73]
Age, Customized [Number; unit: participants]
  < 50 years | 6
  50 - 59 years | 8
  60 - 69 years | 5
  70 - 79 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival Rate
Description: Percentage of participants achieving progression-free survival at 1, 3 and 5 years after the start of protocol therapy, based upon the International Working Group Response Criteria for Non-Hodgkin's Lymphoma (NHL). Progression is defined as a ≥ 50% increase from nadir in the product of the two largest perpendicular diameters (PPD-size) of any previously identified abnormal node, or appearance of any new lesion.
Time Frame: Up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | R-MACLO-IVAM-T
Number analyzed (Participants) | 21
percentage of participants
  1 year progression-free survival | 91 [68 to 98]
  3 year progression-free survival | 78 [51 to 91]
  5-year progression-free survival | 69 [40 to 86]

2. Secondary Outcome: Overall Survival Rate
Description: Percentage of participants who are alive up to five years after receipt of protocol therapy.
Time Frame: Up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | R-MACLO-IVAM-T
Number analyzed (Participants) | 21
percentage of participants
  1-year rate overall survival Rate | 96 [72 to 99]
  2-year overall survival Rate | 96 [72 to 99]
  3-year overall survival rate | 96 [72 to 99]
  4-year overall survival rate | 87 [54 to 96]
  5-year overall survival rate | 87 [54 to 96]

3. Secondary Outcome: Response Rate
Description: Percentage of participants achieving complete response (CR) to protocol therapy according to International Working Group Response Criteria for Non-Hodgkin's Lymphoma (NHL) using the CT imaging method. Patients were classified by best tumor response; CR was defined as normalization of the lactate dehydrogenase (LDH), complete disappearance of disease-related symptoms and lymph nodes, and clearance of lymphoma from involved organs; complete response unconfirmed (CRu) as a residual lymph node greater than 1.5 cm in greatest transverse diameter that had regressed by more than 75% or an indeterminate bone marrow examination; partial response (PR) as greater than 50% reduction in the involved lymph nodes, or disappearance of the involved lymph nodes but persistent bone marrow involvement; relapse/progression as new or increased lymph nodes, organomegaly, or reappearance of bone marrow involvement.
Time Frame: Up to 5 years
Population: Participants who completed at least two cycles of therapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | R-MACLO-IVAM-T
Number analyzed (Participants) | 21
percentage of participants | 100 [83 to 100]

4. Secondary Outcome: Number of Patients Experiencing Adverse Events.
Description: Number of patients experiencing adverse events during the course of protocol therapy.
Time Frame: Up to 5 years
Measure: Number; unit: participants
Groups:
- R-MACLO Cycles: Number of patients experiencing adverse events during the combination Rituximab, Methotrexate, Doxorubicin, Cyclophosphamide and Vincristine (R-MACLO) treatment cycles.
- R-IVAM Cycles: Number of patients experiencing adverse events during the Rituximab, Ifosfamide (and Mesna), Etoposide and Cytarabine (R-IVAM) treatment cycles.
- Thalidomide Therapy: Number of patients experiencing adverse events during Thalidomide maintenance therapy.
Arm/Group | R-MACLO Cycles | R-IVAM Cycles | Thalidomide Therapy
Number analyzed (Participants) | 22 | 22 | 20
participants | 22 | 22 | 19

ADVERSE EVENTS:
Groups:
- R-MACLO Cycles: Adverse Events occurring during the combination Rituximab, Methotrexate, Doxorubicin, Cyclophosphamide and Vincristine (R-MACLO) treatment cycles.
- R-IVAM Cycles: Adverse Events occurring during the Rituximab, Ifosfamide (and Mesna), Etoposide and Cytarabine (R-IVAM) treatment cycles.
- Thalidomide Therapy: Adverse Events occurring during Thalidomide maintenance therapy.
Arm/Group | R-MACLO Cycles | R-IVAM Cycles | Thalidomide Therapy
Serious Adverse Events (participants affected / at risk) | 21/22 | 21/22 | 19/20
Other Adverse Events (participants affected / at risk) | 22/22 | 22/22 | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R-MACLO Cycles (N=22) | R-IVAM Cycles (N=22) | Thalidomide Therapy (N=20)
Neutropenia (Grade 3-4) (Infections and infestations) | 12 (14) | 13 (20) | 7 (7)
Anemia (Grade 3-4) (Metabolism and nutrition disorders) | 7 (7) | 19 (27) | 0 (0)
Thrombocytopenia (Grade 3-4) (Blood and lymphatic system disorders) | 8 (8) | 21 (35) | 0 (0)
Febrile neutropenia (Grade 3-4) (Infections and infestations) | 9 (9) | 20 (20) | 0 (0)
Infection (Grade 3-4) (Infections and infestations) | 5 (5) | 11 (14) | 2 (2)
Bacteremia (Grade 3-4) (Infections and infestations) | 2 (2) | 12 (12) | 0 (0)
Mucositis (Grade 3-4) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Grade 3-4) (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Dyspnea (Grade 3-4) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pleural effusion (Grade 3-4) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Grade 3-4) (General disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral Neuropathy (Grade 3-4) (Nervous system disorders) | 0 (0) | 0 (0) | 8 (8)
Erectile Dysfunction (Grade 3-4) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R-MACLO Cycles (N=22) | R-IVAM Cycles (N=22) | Thalidomide Therapy (N=20)
Neutropenia (Grade 1-2) (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Anemia (Grade 1-2) (Metabolism and nutrition disorders) | 10 (11) | 4 (5) | 0 (0)
Thrombocytopenia (Grade 1-2) (Blood and lymphatic system disorders) | 7 (7) | 0 (0) | 0 (0)
Febrile Neutropenia (Grade 1-2) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0)
Infection (Grade 1-2) (Infections and infestations) | 1 (1) | 5 (5) | 1 (1)
Bacteremia (Grade 1-2) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Grade 1-2) (Metabolism and nutrition disorders) | 10 (11) | 9 (10) | 0 (0)
Hypokalemia (Grade 1-2) (Metabolism and nutrition disorders) | 8 (9) | 11 (14) | 0 (0)
Elevated creatinine (Grade 1-2) (Metabolism and nutrition disorders) | 6 (6) | 4 (4) | 0 (0)
Nausea (Grade 1-2) (General disorders) | 9 (11) | 15 (18) | 0 (0)
Vomiting (Grade 1-2) (General disorders) | 4 (4) | 10 (10) | 0 (0)
Mucositis (Grade 1-2) (Infections and infestations) | 11 (13) | 8 (9) | 0 (0)
Diarrhea (Grade 1-2) (Gastrointestinal disorders) | 5 (5) | 6 (6) | 0 (0)
Constipation (Grade 1-2) (Gastrointestinal disorders) | 6 (6) | 5 (7) | 7 (7)
Dyspnea (Grade 1-2) (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5) | 0 (0)
Edema (Grade 1-2) (General disorders) | 6 (6) | 3 (3) | 4 (4)
Pleural Effusion (Grade 1-2) (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
Headache (Grade 1-2) (General disorders) | 9 (10) | 4 (6) | 0 (0)
Dizziness (Grade 1-2) (General disorders) | 2 (3) | 4 (5) | 2 (2)
Rash (Grade 1-2) (Infections and infestations) | 5 (5) | 8 (9) | 0 (0)
Somnolence (Grade 1-2) (General disorders) | 0 (0) | 0 (0) | 3 (3)
Peripheral Neuropathy (Grade 1-2) (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Erectile Dysfunction (Grade 1-2) (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Grade 1-2) (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes